CLINICAL TRIAL: NCT01779505
Title: A Randomized, Open-Label, Multi-Arm, Dose Escalation, Phase 1a Trial Assessing the Safety, Tolerability, and Immunogenicity of GI-13020; an Inactivated Recombinant Saccharomyces Cerevisiae Expressing Hepatitis B Virus X, Surface and Core Antigens, at Various Dose Levels and Regimens in Healthy Adults.
Brief Title: A Phase 1a Trial Assessing the Safety, Tolerability, and Immunogenicity of GS-4774 (GI-13020) at Various Dose Levels and Regimens in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GI-13020-01
Record Dates: First submitted 2013-01-24; First posted 2013-01-30 (Estimated); Last update posted 2014-01-08 (Estimated); Status verified 2014-01

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- GS-4774 at 10 yeast units (YU) (Experimental): 10 YU of GS-4774 given either weekly or monthly
  Interventions: Biological: GS-4774
- GS-4774 at 40 YU (Experimental): 40 YU of GS-4774 given either weekly or monthly
  Interventions: Biological: GS-4774
- GS-4774 at 80YU (Experimental): 80 YU of GS-4774 given either weekly or monthly
  Interventions: Biological: GS-4774

INTERVENTIONS:
Biological: GS-4774 — GS-4774 is a recombinant yeast-based biological product engineered to express HBV antigens. The product is a heat-killed yeast (S. cerevisiae) containing a chimera of HBV X, Score, and Core antigens.
  Other Names: GI-13020

SUMMARY:
This trial will be test the safety, tolerability, and immunogenicity of GS-4774 (GI-13020) in various doses and dosing regimens in healthy adults at one center in the US. Subjects will be enrolled into 3 arms using a dose escalation scheme and randomized into one of two dosing regimen cohorts. There will be 10 subjects per arm/cohort (total of 60 subjects to achieve 48 evaluable subjects enrolled), with study completion in 9-12 months.

DETAILED DESCRIPTION:
HBV specific T cell responses have been shown to have a positive association with infection status in patients with chronic HBV, with the weakest T cell responses in patients with untreated chronic active infection and the strongest T cell responses in patients who have achieved seroconversion or cure (4). We have generated a Tarmogen expressing well conserved regions of the HBV X, S, and core antigens (GS-4774). GS-4774 is immunogenic in murine models and has also been used to stimulate human immune cell samples ex vivo to elicit HBV specific T cell responses which could predict the immune responses in patients dosed with GS-4774. GS-4774 will be evaluated in this healthy volunteer study to assess its safety, tolerability, and ability to elicit HBV specific T cell responses. In the future GS-4774 could be used in combination with HBV antivirals, such as tenofovir disoproxil fumarate, in an attempt to improve HBsAg seroconversion (cure) rates in patients with chronic HBV infection.

ELIGIBILITY:
Inclusion Criteria:

* Signed, written, informed consent from the subject before any study-specific procedures are performed
* Free of obvious health problems as established by medical history and clinical examination before entering into the study
* If female, negative pregnancy test and for women of childbearing potential willingness to use reliable method of birth control during the study and for 30 days after the last dose of study medication
* Male or female aged ≥ 18 years at the time of first dose
* Negative scratch test (immediate hypersensitivity, immunoglobulin E (IgE) mediated) to S. cerevisiae

Exclusion Criteria:

* Hospitalization in the last 6 months
* No medicine adjustments in the last 6 months
* History of anaphylaxis from any cause
* History of hepatitis B virus (HBV) infection as evidenced by detection of HBV Surface and Core antigens
* History of vaccination with HBV prophylactic vaccine or positive for antibody to HBV Surface and Core antigens
* Known exposure to HBV within the past 6 weeks
* Increased alpha fetoprotein (AFP) at screening
* History of hepatitis C virus (HCV) infection or positive HCV antibody, Herpes zoster, shingles or any other chronic viral infection
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests
* Known history of HIV infection or positive HIV antibody test at screening
* History of demyelinating disease such as Guillain-Barre Syndrome
* History of Bell's Palsy
* Immunosuppression as a result of underlying illness or treatment
* History of cancer within the last 5 years with the exception of localized basal or squamous cell carcinoma or Stage 1A cervical cancer
* History of Crohn's disease or ulcerative colitis
* History of autoimmune disease
* History of organ transplantation
* Concurrent and chronic therapy with immunosuppressive drugs including systemic corticosteroids
* Receipt of investigational drugs or vaccines within 30 days or 5 half lives, whichever is longer, prior to first injection with the study drug
* Receipt of immunoglobulin or other blood products within 3 months prior to enrollment
* Receipt of allergy shots within the preceding 7 days or expected to receive allergy shots during the study and 7 days following completion of study
* Receipt of biologics
* Negative histamine response on scratch test at screening
* High risk for noncompliance with the protocol
* Alcohol and/or IV drug abuse within the past year
* Positive urine drug test at screen visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-01; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Safety of GS-4774 at various doses | 6 months
  Frequency of serious adverse events Frequency and severity of common non-serious adverse events Frequency of discontinuations of therapy due to adverse events Common laboratory assessments (chemistry, hematology, urinalysis) Dose Limiting Toxicities

SECONDARY OUTCOMES:
Immunogenicity of various doses and dosing regimens of GS-4774 | 6 months
  Frequency and magnitude of antigen specific immune responses by enzyme-linked immunosorbent spot (ELISpot) assay for cytokine production, to include interferon gamma (IFNγ) Frequency and magnitude of antigen specific immune responses by lymphocyte proliferation assay (LPA) Frequency and magnitude of anti-Saccharomyces cerevisiae antibody (ASCA) responses Pentamer staining for HBV specific T cells Frequency of regulatory T cells (Treg) responses

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion, Phoenix, Arizona, United States

REFERENCES:
- [Derived] Gaggar A, Coeshott C, Apelian D, Rodell T, Armstrong BR, Shen G, Subramanian GM, McHutchison JG. Safety, tolerability and immunogenicity of GS-4774, a hepatitis B virus-specific therapeutic vaccine, in healthy subjects: a randomized study. Vaccine. 2014 Sep 3;32(39):4925-31. doi: 10.1016/j.vaccine.2014.07.027. Epub 2014 Jul 18. PMID 25045824